CLINICAL TRIAL: NCT05027971
Title: Flexiva Pulse Laser Fiber Post-Market Patient Registry
Brief Title: Flexiva Pulse Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 92704912
Record Dates: First submitted 2021-08-06; First posted 2021-08-31 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Urinary Calculi; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Urinary Calculi; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Lithotripsy Cohort: Subjects in this cohort will undergo lithotripsy procedure for the treatment of urinary calculi.
  Interventions: Device: Flexiva Pulse High Power Single-Use Laser Fibers
- Benign Prostatic Hyperplasia (BPH) Cohort: Subjects in this cohort will undergo Holmium Laser Enucleation of the Prostate (HoLEP) procedure for the treatment of BPH.
  Interventions: Device: Flexiva Pulse High Power Single-Use Laser Fibers

INTERVENTIONS:
Device: Flexiva Pulse High Power Single-Use Laser Fibers — Flexiva Pulse High Power Single-Use Laser Fibers are intended to be used as a device that transmits Ho:YAG laser energy from cleared laser consoles to urological anatomy.

SUMMARY:
To obtain post-market safety and efficacy data for FlexivaTM Pulse High Power Single-Use Laser Fibers during lithotripsy and soft tissue procedure of holmium laser enucleation of the prostate (HoLEP).

DETAILED DESCRIPTION:
Multi-center, open label, prospective study to document on-going post-market safety and performance of Flexiva Pulse High Power Single-Use Laser Fibers.

All subjects meeting the enrollment criteria, signing the consent and undergoing the lithotripsy/HoLEP procedure with the study device(s) will be followed: up to 2 months (60 days) post-discharge from final holmium laser lithotripsy procedure for subjects in the lithotripsy cohort or up to 6 months (180 days + 60 days) post discharge from HoLEP procedure for subjects in the Benign Prostatic Hyperplasia (BPH) cohort.

ELIGIBILITY:
Inclusion Criteria:

For Lithotripsy cohort:

1. Subject is undergoing treatment for urinary calculi
2. Subject is willing and able to return for all follow-up visits

For BPH cohort:

1. Subject is ≥ 40 years of age
2. Subject with a diagnosis of benign prostatic hyperplasia (BPH) with lower urinary tract symptoms
3. IPSS (International Prostate Symptom Score) ≥ 12
4. Qmax (Peak Flow Rate) ≤ 15 mL/s
5. Subject is willing and able to return for all follow-up visits

Exclusion Criteria:

For Lithotripsy cohort:

1. Subject has uncontrolled bleeding disorders and coagulopathy
2. Subject has untreated urinary tract infection (UTI)
3. Subject requires simultaneous HoLEP procedure

For BPH cohort:

1. Subject has a diagnosis of bladder cancer
2. Subject has a diagnosis of prostate cancer
3. Subject with prostate-specific antigen (PSA) ˃ 10 ng/mL suggestive of prostate cancer is not eligible unless patient has concomitant negative prostate biopsy
4. Subject has acute prostatitis, a prostate abscess, or neurogenic bladder
5. Subject has urethral stricture disorder
6. Subject has uncontrolled bleeding disorders and coagulopathy
7. Subject has untreated urinary tract infection (UTI)
8. Subject requires simultaneous upper urinary calculi lithotripsy procedure (not applicable to bladder calculi)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 200 subjects will be enrolled and treated for lithotripsy of urinary calculi and BPH indications. There will be about 100 subjects enrolled in the lithotripsy cohort and 100 subjects enrolled in the BPH cohort.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinic Pheonix, Phoenix, Arizona
  - University of Miami, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Lehigh Valley Hospital, Allentown, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were considered enrolled in the study after signing and dating the informed consent form and after the lithotripsy/HoLEP procedure was attempted. There was a total of 209 subjects consented and 8 subjects were exited prior to procedure, resulting in a total of 201 subjects enrolled.
Period: Overall Study
Arm/Group | Lithotripsy Cohort | Benign Prostatic Hyperplasia (BPH) Cohort
Started | 105 | 104
Completed | 97 | 95
Not Completed | 8 | 9
Not completed — Physician Decision | 7 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Non-study fiber used. | 0 | 1
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: Five subjects exited prior to procedure initiation in the Lithotripsy Cohort and 3 subjects exited prior to procedure initiation in the HoLEP cohort. One subject in the Lithotripsy Cohort was withdrawn by investigator after procedure was initiated and no stones were present for use of the Flexiva Pulse Laser Fiber.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithotripsy Cohort | Benign Prostatic Hyperplasia (BPH) Cohort | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  18-64 years | 76 | 37 | 113
  ≥65 years | 23 | 64 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 0 | 46
  Male | 53 | 101 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 24 | 66
  Not Hispanic or Latino | 52 | 73 | 125
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 9 | 11
  White | 87 | 83 | 170
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 101 | 200

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Serious Adverse Device Effects - Primary Safety Endpoint
Description: The primary safety endpoint is the occurrence of Serious Adverse Device Effects (SADE) related to Flexiva Pulse Laser Fibers during lithotripsy procedures.
Time Frame: Up to 60 days of follow-up for Lithotripsy Cohort
Population: The primary analysis was performed for the Intent to Treat (ITT) population. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study and had the lithotripsy procedure attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Lithotripsy Cohort
Number analyzed (Participants) | 100
Participants | 2
Statistical Analysis 1: Comparison: Lithotripsy Cohort; Test type: Other; Proportion by cohort = .02, 95% CI 2-sided [.002 to .07]

2. Primary Outcome: Occurrence of Serious Adverse Device Effects - Primary Safety Endpoint
Description: The primary safety endpoint is the occurrence of Serious Adverse Device Effects (SADE) related to Flexiva Pulse Laser Fibers during HoLEP procedures.
Time Frame: Up to 240 days of follow-up for BPH Cohort.
Population: The primary analysis was performed for the Intent to Treat (ITT) population. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study and had the HoLEP procedure attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Prostatic Hyperplasia (BPH) Cohort
Number analyzed (Participants) | 101
Participants | 3
Statistical Analysis 1: Comparison: Benign Prostatic Hyperplasia (BPH) Cohort; Test type: Other; Proportion by cohort = .03, 95% CI 2-sided [.006 to .084]

3. Primary Outcome: Stone Free Rates - Primary Efficacy Endpoint 1
Description: In lithotripsy procedures: Stone clearance assessed by stone free rates (SFR) at the 1 month follow-up. Stone free was defined as clinically nonsignificant, non-obstructive residual fragments of ≤ 3 mm, asymptomatic, and no auxiliary procedures performed between the final Flexiva Pulse holmium laser lithotripsy procedure and the 1-month follow-up.
Time Frame: 1 month follow-up
Population: The proportion of subjects who achieved stone clearance at 1 month follow-up post lithotripsy procedure was calculated. The analysis used all available cases and the last available visit data was analyzed if multiple post operative visits occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Lithotripsy Cohort
Number analyzed (Participants) | 81
Participants | 54
Statistical Analysis 1: Comparison: Lithotripsy Cohort; Test type: Other; Proportion by cohort = .667, 95% CI 2-sided [.553 to .768]

4. Primary Outcome: Change in BPH Symptoms - Primary Efficacy Endpoint 2
Description: In HoLEP procedures: Improvement in BPH symptoms from baseline as measured by favorable change (decrease) in International Prostate Symptom Score (IPSS) at 3 month follow-up, on a scale of 0 to 35.
Time Frame: 3 month follow-up
Population: Change in IPSS total score in BPH subjects from baseline to 3 month post procedure was analyzed. If multiple IPSS scores were collected during the analysis window, only the last IPSS score collected in the window was counted. Visits that occurred from 60 days through 150 days post-operative were considered as 3-month visits. IPSS cannot be obtained in catheterized subjects; 30 subjects had catheters at baseline. 57 subjects had data at both baseline and 3 months post procedure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benign Prostatic Hyperplasia (BPH) Cohort
Number analyzed (Participants) | 57
score on a scale | -15.8 (6.1)
Statistical Analysis 1: Comparison: Benign Prostatic Hyperplasia (BPH) Cohort; Test type: Other; Mean Difference (Final Values) = -15.8, 95% CI 2-sided [-17.4 to -14.2]

5. Secondary Outcome: Procedure Related AEs and/or ADEs - Secondary Safety Endpoint
Description: Procedure related adverse events and/or adverse device effects related to Flexiva Pulse Laser Fibers, including but not limited to:
  * Perforation: For Lithotripsy procedures: anywhere in urinary tract.
  * Hemorrhage resulting in blood loss of ≥ 500mL
  * Burn
Time Frame: Up to 60 days of follow-up for Lithotripsy Cohort
Population: The analysis was performed for the Intent to Treat (ITT) population. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study and had the lithotripsy procedure attempted. There were no reports of perforations, hemorrhages, or burns in the Lithotripsy cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Lithotripsy Cohort
Number analyzed (Participants) | 100
Participants | 6

6. Secondary Outcome: Procedure Related AEs and/or ADEs - Secondary Safety Endpoint
Description: Procedure related adverse events and/or adverse device effects related to Flexiva Pulse Laser Fibers, including but not limited to:
  * Perforation: For HoLEP procedures: in prostate capsule, bladder, and/or urethra
  * Hemorrhage resulting in blood loss of ≥ 500mL
  * Burn
Time Frame: Up to 240 days of follow-up for BPH Cohort.
Population: The analysis was performed for the Intent to Treat (ITT) population. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study and had the lithotripsy procedure attempted. There were no reports of perforations or burns in the BPH cohort; 2 hemorrhages occurred in the ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Prostatic Hyperplasia (BPH) Cohort
Number analyzed (Participants) | 101
Participants | 31

7. Secondary Outcome: Ability of Fiber to Deliver Energy - Secondary Efficacy Endpoint 1
Description: For Lithotripsy procedures:
  • Ability of the laser fiber to deliver energy as measured by whether or not the Lithotripsy procedure was successfully completed as indicated. Tool used will be a yes or no question on the case report form.
Time Frame: Through lithotripsy procedure completion, up to 1 day.
Population: Statistics are based on the number of Flexiva Pulse fibers used in all subjects for which data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Lithotripsy Cohort
Number analyzed (Participants) | 98
Participants | 98
Statistical Analysis 1: Comparison: Lithotripsy Cohort; Test type: Other; Proportion by cohort = 1, 95% CI 2-sided [.963 to 1]

8. Secondary Outcome: Ability of Fiber to Deliver Energy - Secondary Efficacy Endpoint 2
Description: For HoLEP procedures:
  Ability of the laser fiber to deliver energy as measured by whether or not the HoLEP procedure was successfully completed as indicated. Tool used will be a yes or no question on the case report form.
Time Frame: Through HoLEP procedure completion, up to 1 day.
Population: Statistics are based on the number of Flexiva Pulse fibers used in all subjects for which data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Prostatic Hyperplasia (BPH) Cohort
Number analyzed (Participants) | 99
Participants | 99
Statistical Analysis 1: Comparison: Benign Prostatic Hyperplasia (BPH) Cohort; Test type: Other; Proportion by cohort = 1, 95% CI 2-sided [.963 to 1]

9. Secondary Outcome: Fiber and Scope Compatibility - Secondary Efficacy Endpoint 1
Description: For Lithotripsy procedures:
  • Compatibility of the laser fiber with endoscope as measured by whether or not the laser fiber is compatible with the endoscope used in the index procedure, including successful passage and maneuverability without fracture. Tool used will be a yes or no question on the case report form.
Time Frame: Through lithotripsy procedure completion, up to 1 day.
Population: Statistics are based on the number of Flexiva Pulse fibers used in all subjects for which data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Lithotripsy Cohort
Number analyzed (Participants) | 98
Participants | 98
Statistical Analysis 1: Comparison: Lithotripsy Cohort; Test type: Other; Proportion by cohort = 1, 95% CI 2-sided [.963 to 1]

10. Secondary Outcome: Fiber and Scope Compatibility - Secondary Efficacy Endpoint 2
Description: For HoLEP procedures:
  • Compatibility of the laser fiber with endoscope as measured by whether or not the laser fiber is compatible with the endoscope used in the index procedure, including successful passage and maneuverability without fracture. Tool used will be a yes or no question on the case report form.
Time Frame: Through HoLEP procedure completion, up to 1 day.
Population: Statistics are based on the number of Flexiva Pulse fibers used in all subjects for which data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Prostatic Hyperplasia (BPH) Cohort
Number analyzed (Participants) | 99
Participants | 88
Statistical Analysis 1: Comparison: Benign Prostatic Hyperplasia (BPH) Cohort; Test type: Other; Proportion by cohort = .889, 95% CI 2-sided [.810 to .943]

11. Secondary Outcome: Change in Uroflowmetry - Secondary Efficacy Endpoint 2
Description: For HoLEP procedures:
  • Improvement in uroflowmetry from baseline as measured by change (increase) in maximum urinary flow rate (Qmax) at 3-month follow-up
Time Frame: Up to 3 month follow-up
Population: The analysis was performed for the Intent to Treat (ITT) population where Qmax was available at baseline and at 3 months post procedure. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study and had the HoLEP procedure attempted. Qmax was available for 58 subjects at both timepoints.
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Benign Prostatic Hyperplasia (BPH) Cohort
Number analyzed (Participants) | 58
mL/s | 15.0 (13.9)
Statistical Analysis 1: Comparison: Benign Prostatic Hyperplasia (BPH) Cohort; Test type: Other; Mean Difference (Final Values) = 15.0, 95% CI 2-sided [11.3 to 18.6]

12. Secondary Outcome: Change in Quality of Life - Secondary Efficacy Endpoint 2
Description: For HoLEP procedures:
  Improvement in Quality of Life (QoL) from baseline as measured by favorable change (decrease) in International Prostate Symptom Score (IPSS) at 3-month follow-up, on a scale of 0 to 6.
Time Frame: Up to 3 month follow-up
Population: The primary analysis was performed for the Intent to Treat (ITT) population where the IPSS QoL score was available at baseline and at 3 months post procedure. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study and had the HoLEP procedure attempted. IPSS QoL score was available for 41 subjects at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benign Prostatic Hyperplasia (BPH) Cohort
Number analyzed (Participants) | 41
score on a scale | -3.4 (1.6)
Statistical Analysis 1: Comparison: Benign Prostatic Hyperplasia (BPH) Cohort; Test type: Other; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-3.9 to -2.9]

13. Secondary Outcome: Hemostasis - Secondary Efficacy Endpoint 2
Description: For HoLEP procedures:
  • Hemostasis measured by ability to coagulate during HoLEP procedure. Tool used will be a yes or no question on the case report form.
Time Frame: Through HoLEP procedure completion, up to 1 day.
Population: The analysis was performed for the Intent to Treat (ITT) population. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study and had the HoLEP procedure attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Prostatic Hyperplasia (BPH) Cohort
Number analyzed (Participants) | 99
Participants | 99
Statistical Analysis 1: Comparison: Benign Prostatic Hyperplasia (BPH) Cohort; Test type: Other; Proportion by cohort = 1, 95% CI 2-sided [.963 to 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of index procedure to end of the study for each subject enrolled (up to 60 days post lithotripsy procedure and up to 240 days post HoLEP procedure).
Description: AE reporting included: Serious Adverse Device Effects, Procedure Related Serious Adverse Events, Fatal Serious Adverse Events, Adverse Device Effects, and Procedure Related Adverse Events
Arm/Group | Lithotripsy Cohort | Benign Prostatic Hyperplasia (BPH) Cohort
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/101
Serious Adverse Events (participants affected / at risk) | 2/100 | 6/101
Other Adverse Events (participants affected / at risk) | 4/100 | 27/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithotripsy Cohort (N=100) | Benign Prostatic Hyperplasia (BPH) Cohort (N=101)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 2 (3)
Bladder Stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatic Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithotripsy Cohort (N=100) | Benign Prostatic Hyperplasia (BPH) Cohort (N=101)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Pyelitis (Infections and infestations) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 1 (1) | 12 (12)
Haematuria (Renal and urinary disorders) | 0 (0) | 7 (7)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 5 (5)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder Spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pelvic Discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Device Occlusion (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT05027971/Prot_SAP_000.pdf